CLINICAL TRIAL: NCT01102751
Title: Effects Of Vitamin D Replacement Therapy on Serum FGF-23 Concentrations in Vitamin D Deficient Women In Short Term
Brief Title: Serum FGF-23 and Vitamin D Deficiency
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Other Study IDs: Istanbul University; Research Fund (Other: 573/05052006)
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2009-08

CONDITIONS: Osteomalacia
Keywords: fibroblast growth factor 23; Osteomalacia; vitamin D
MeSH Terms: conditions — Osteomalacia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Vitamin D deficient females: (n =18, mean age 29.1±9.9 yrs)
- vitamin D sufficient healthy females: (control group; n = 19, mean age 28.5±5.2 yrs)
- genetically-determined hypophosphatemic rahitis: (n=13, mean age 26.5±15.1 yrs)

SUMMARY:
We aimed to determine the effect of vitamin D replacement therapy on serum FGF-23 concentrations in vitamin D deficient women and to compare the FGF-23 concentrations of vitamin D deficient patients with healthy subjects and patients with genetically-determined hypophosphatemic rickets.

DETAILED DESCRIPTION:
Study group was composed of vitamin D deficient females (n =18, mean age 29.1±9.9 yrs), vitamin D sufficient healthy females (control group; n = 19, mean age 28.5±5.2 yrs) and patients with genetically-determined hypophosphatemic rickets (n=13, mean age 26.5±15.1 yrs). Groups were compared for serum FGF-23, 1,25 dihydroxy vitamin D3, calcium, phosphate, bone turnover markers, intact parathyroid hormone and urinary excretion of calcium and phosphate. Vitamin D deficient group was re-evaluated after a standard treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Serum 25OHD Vitamin <30 ng/mL for group 1
* Serum 25OHD Vitamin >30 ng/mL for control group

Exclusion Criteria:

* Receiving medication(s) affecting bone metabolism
* History of gastrointestinal disease and malabsorption
* History of renal and liver disease

Ages: 9 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Group 1: Eighteen premenopausal female patients with a diagnosis of vitamin D deficient osteomalacia were included in this group. Vitamin D deficiency was diagnosed according to the serum 25 hydroxy vitamin D3 (25OHD) concentrations (< 30 ng/mL). Reasons for vitamin D deficiency were verified as insufficient exposure to sunlight, frequent parturition and prolonged lactation. All of these patients received a standard treatment regimen; oral Vitamin D3 150 000 IU once for all and subsequently 880 IU D3 and 1000 mg calcium carbonate for six weeks. This group was also evaluated after replacement therapy at sixth week.
  Group 2: Nineteen healthy premenopausal women who had normal levels of serum 25OHD Vitamin (>30 ng/mL) composed the control group.
  Group 3: Thirteen hypophosphatemic rickets (3 autosomal dominant and 10 X-linked; 9 female and 4 male) were included in this group.
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Department of Internal Medicine, Division of Endocrinology and Metabolism, Istanbul, Turkey (Türkiye)